CLINICAL TRIAL: NCT03424720
Title: Comparative Analysis of Phase Lag Entropy (PLE) and Bispectral Index (BIS) as an Anesthetic Depth Indicator in Patients Undergoing Otopharyngeal Surgery With Facial Nerve Integrity Monitoring
Brief Title: Comparative Analysis of Phase Lag Entropy (PLE) and Bispectral Index (BIS) as an Anesthetic Depth Indicator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Kyung Mi Kim, Staff, Department of Anesthesiology and pain Medicine, Principal Investigator, Assistant Professor., Hallym University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3-2017-10047988
Record Dates: First submitted 2018-01-17; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: General Anesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparison of PLE and BIS (Experimental): Investigators assess PLE and BIS values as indicators of the depth of anesthesia during induction and emergence of anesthesia and facial nerve integrity monitoring
  Interventions: Device: PLE and BIS

INTERVENTIONS:
Device: PLE and BIS — Investigators attach the PLE and BIS sensors on the forehead of the patients undergoing facial nerve integrity monitoring during general anesthesia using total intravenous anesthetics

SUMMARY:
The aim of this comparative analysis is to evaluate the reliability of PLE value as an anesthetic depth indicator

DETAILED DESCRIPTION:
1. To evaluate the reliability of PLE value as an anesthetic depth indicator, the investigators compare PLE value with BIS score during induction and emergence of general anesthesia using propofol target controlled infusion.
2. In addition, the investigators verify whether or not the facial nerve integrity monitoring affects the efficacy for PLE and BIS values as an anesthetic depth indicator.

ELIGIBILITY:
Inclusion Criteria:

* Patients who scheduled for otopharyngeal surgery under facial nerve integrity monitoring requiring general anesthesia and American Society of Anesthesiology (ASA) physical status 1 or 2

Exclusion Criteria:

* Patient who has been taken anticonvulsant agents, sedatives, and hypnotics
* Patient who has central nerve system disease, neurological disorder
* Patient with hypersensitivity to anesthetics

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-08-02 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
PLE value during induction and emergence of general anesthesia | Through study completion, an average of fifteen months
  Investigators measure the PLE value as an anesthetic depth indicator before the injection of propofol, at the time point of no response to verbal command, before and after intubation, and at the time point of response to verbal command during emergence of anesthesia.
  The PLE value will be reported in a score ranging from 0 (burst suppression or deep sedated) to 100 (full awake).

SECONDARY OUTCOMES:
BIS value during induction and emergence of general anesthesia | Through study completion, an average of fifteen months
  Investigators measure the BIS value as an anesthetic depth indicator before the injection of propofol, at the time point of no response to verbal command, before and after intubation, and at the time point of response to verbal command during emergence of anesthesia.
  The BIS value will be reported in a score ranging from 0 (burst suppression or deep sedated) to 100 (full awake).
PLE value during facial nerve integrity monitoring | Through study completion, an average of fifteen months
  Investigators measure the PLE value at the time points of facial nerve integrity monitoring.
  The PLE value will be reported in a score ranging from 0 (burst suppression or deep sedated) to 100 (full awake).
BIS value during facial nerve integrity monitoring | Through study completion, an average of fifteen months
  Investigators measure the BIS value at the time points of facial nerve integrity monitoring.
  The BIS value will be reported in a score ranging from 0 (burst suppression or deep sedated) to 100 (full awake).

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Mi Kim, Ph.D., Principal Investigator — Department of Anesthesiology and Pain Medicine
Locations (1):
- Hallym University Medical Center, Anyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No